CLINICAL TRIAL: NCT03762044
Title: New Therapeutic Approach in Upper Limb Lymphedema Secondary to Breast Cancer: Activity-oriented Proprioceptive Antiedema Therapy (TAPA). A Randomized Controlled Therapy
Brief Title: New Therapeutic Approach in Upper Limb Lymphedema Secondary to Breast Cancer: Activity-oriented Proprioceptive Antiedema Therapy (TAPA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Reina Sofia de Cordoba (Other Government)
Responsible Party: Principal Investigator, Antonio José Jiménez Vílchez, Physical Medicine & Rehabilitation Hospital Resident, Hospital Universitario Reina Sofia de Cordoba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Lymphedema Rehabilitation
Record Dates: First submitted 2018-11-23; First posted 2018-12-03 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Breast Cancer Lymphedema; Post-Mastectomy Secondary Lymphedema
Keywords: Breast Cancer; Breast Cancer Lymphedema; Post-Mastectomy Secondary Lymphedema; Occupational Therapy; Proprioceptive Neuromuscular Facilitation; Neural Mobilization
MeSH Terms: conditions — Breast Cancer Lymphedema; Breast Neoplasms | interventions — tapasin

STUDY DESIGN:
Intervention Model Description: After proposing to the subjects the enrollment to the study and once they accept, they will be randomly allocated to experimental TAPA treatment group or standard CDT treatment. They will be assessed 1 to 3 days before and after completing the treatment. It will be consists in a total of 10 sessions of 30 minutes of treatment, twice per week in a total 5 weeks period.
Who Masked: Investigator, Outcomes Assessor
Masking Description: In order to masking, investigator who assess the subject before and after the treatment will not know which group the subjects belong, and so the biostatistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Activity-oriented Proprioceptive Antiedema Therapy (TAPA) (Experimental): 10 sessions of 30 minutes, twice a week in a total 5 week period of Activity-oriented Proprioceptive Antiedema Therapy (TAPA in Spanish)
  Interventions: Other: Activity-oriented Proprioceptive Antiedema Therapy (TAPA)
- Complete Decongestive Therapy (CDT) (Active Comparator): 10 sessions of 30 minutes, twice a week in a total 5 week period of complete decongestive therapy (CDT).
  Interventions: Other: Complete Decongestive Therapy (CDT)

INTERVENTIONS:
Other: Activity-oriented Proprioceptive Antiedema Therapy (TAPA) — * Health education / patient empowerment.
  * Neurodynamic activities oriented to ADL.
  * Proprioceptive neuromuscular facilitation exercises oriented to ADL.
  * Self-adherent self-adhesive antiedema of low compression.
  Arms: Activity-oriented Proprioceptive Antiedema Therapy (TAPA)
Other: Complete Decongestive Therapy (CDT) — * Skin care.
  * Kinesitherapy
  * Manual lymphatic drainage (MLD)
  * Multilayer bandage.
  The maintenance phase is based on self-care and the use of compression garments.
  Arms: Complete Decongestive Therapy (CDT)

SUMMARY:
This study evaluates the effectiveness of an experimental proposal therapy for upper limb lymphedema secondary to breast called Activity-oriented proprioceptive antiedema therapy (TAPA) facing the consensual gold standard treatment, the complete decongestive therapy. TAPA consists in:

* Health education / patient empowerment.
* Neurodynamic activities oriented to Activities of Daily Living (ADL).
* Proprioceptive neuromuscular facilitation exercises oriented to ADL.
* Self-adherent self-adhesive antiedema of low compression.

Half of patients will receive TAPA treatment while the other half will receive CDT standard treatment.

DETAILED DESCRIPTION:
Lymphedema is defined as the abnormal accumulation of tissue proteins, which is accompanied of edema and chronic inflammation of a limb, so post-mastectomy lymphedema is one of the most serious sequelae of Breast Cancer (BC) that affects the quality of life of women operated for breast cancer. Its incidence is approximately between 6 and 30% of patients and its prevalence varies between 15-20%. It is considered a process without spontaneous resolution that involves the application of a palliative therapy conservative for life, with preventive measures to reduce it and prevent complications and an expected increase in the number of patients with lymphedema in the next years

Changes in work performance resulting from lymphedema vary from minor temporary changes to significant difficulties in the ADL, depending on the chronicity and severity of the affectation. It could affect physical components and psychological, as well as social and economic environment. In these limitations on activities and / or restrictions of participation, the Occupational Therapists (OT) provide a unique approach, since they are professionals specifically enabled for the use of the therapeutic potential of the activity and graduation of its control parameters in favor of the best occupational performance possible of the person. Furthermore, there are some research that support the inclusion of OT in the cancer rehabilitation and reveal a significant need for more research to explore ways in which the OT favorably influences the results of the cancer survivors.

The anamnesis, clinical exploration and complementary studies if necessary, allow us confirm the diagnosis of lymphedema, stage, possibilities of progression and approach the most indicated therapeutic in each case.

The conservative therapeutic of upper limb lymphoedema secondary to breast cancer plan includes preventive exercises and lifestyle habits, complete decongestive therapy (CDT) and compression garments.

The CDT comprises a series of measures, a first intensive phase consists of:

* Skin care.
* Kinesitherapy
* Manual lymphatic drainage (MLD)
* Multilayer bandage. The maintenance phase is based on self-care and the use of compression garments.

Despite the consensus of the experts in the evidence of decongestive therapy in lymphedema, there is still a lack of evidence to inform the optimal doses of treatment and the level of evidence about its efficacy in the treatment of lymphedema is only moderately strong, due to the scarcity of randomized trials with control group, well interventions controlled, accurate measures of volume, mobility or function and quality of life.

Likewise, the prescription of compression garments for lymphoedema is very varied and it may be due to the lack of underlying evidence to inform about the treatment. The evidence also suggests that the comprehensiveness and effectiveness of rehabilitation post-operative BC should also consider the self-control (empowerment) of patients, approaches to redesign the lifestyle and incorporate aspects of the promotion of health.

On the other hand, there are studies that confirm that women with lymphedema and pain after BC may present alterations in neural mechanosensitivity, neuropathic pain, as a result of nerve compression or peripheral neuropathy induced by chemotherapy and that it is worth conducting a clinical trial to evaluate the techniques of Neural mobilization (NM) oriented to the functionality of upper extremities, supporting the clinical mechanism of NM in the reduction of intraneural edema.

Published research suggests incorporating proprioceptive neuromuscular facilitation (PNF) with the traditional NM method, to facilitate the process of treatment for patients with lymphoedema, because it induces powerful synergistic effects on the volume of edema, range of motion (ROM) of the shoulder, pain and depression. That treatment independently or in combination with laser also improves these variables and even the speed of blood circulation in the armpit. Furthermore, in a study in which bandaging could not be used and CDT was combined with PNF and respiration, reducing lymphedema and improving ROM too, which could improve performance of activities, level of participation and, therefore, quality of life.

There are research supporting use of Coban®3M bandage as early start of pressotherapy in the rehabilitation treatment of lymphedema to reduce prolonged edema (agent cause of multiple complications and functional loss), we consider the possibility of testing the efficacy of a bandage with similar characteristics, in terms of elasticity and self-adherence, more economical, applying it from distal to proximal, with a low level of compression, in order to provide proprioceptive information, but avoiding compressive syndrome, reducing pain and edema and improving the performance of ADL through the practice of them. It consists in only two thin layers and it is fast (10 minutes) and simple placement (can be self-administered by the patient and / or caregiver), improving cost- effectiveness of treatments combined with three other techniques whose evidence has been previously reviewed. We have agreed to call this therapy we propose in this study Activity-oriented Proprioceptive Antiedema Therapy (TAPA in Spanish):

* Health education / patient empowerment.
* Neurodynamic activities oriented to ADL.
* Proprioceptive neuromuscular facilitation exercises oriented to ADL.
* Self-adherent self-adhesive antiedema of low compression.

Given the consensus of the CDT as a gold standard treatment in lymphedema, we consider that our experimental treatment TAPA should make the comparison with it. So, half of patients will receive TAPA treatment while the other half will receive CDT standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Upper limb lymphedema secondary to breast cancer grade I and II, according to the Working Group of the XI International Lymphology Congress

Exclusion Criteria:

* Upper limb lymphedema secondary to breast cancer grade 0 and III, according to the Working Group of the XI International Lymphology Congress

Ages: 14 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — It consists in women with upper limb lymphedema secondary to breast cancer
Enrollment: 51 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Volume | Baseline and 5 weeks
  Volume of the upper limb lymphedema using the Kuhnke formula (Vol=(C1^2+C2^2+...Cn^2)/π). It allows you to assess the volume difference between the affected limb and the healthy one. According to the Working Group of the XI International Lymphology Congress, lymphedema are classified in grade I (mild) ( 10-25% difference), grade II (moderate) (26-50% difference) and grade III (severe) (>51% difference).
Circometry | Baseline and 5 weeks
  Perimeter of upper limb lymphedema using a measuring tape in seven spots: Metacarpophalangeal, 5 and 10cm over radial styloid, 5cm under lateral epicondyle and 5, 10 and 15cm over lateral epicondyle. It is significative when there is a 2cm difference between the healthy and affected limb.

SECONDARY OUTCOMES:
Quick Disabilities of the Arm, Shoulder and Hand (Quick DASH) | Baseline and 5 weeks
  Upper limp function for development of activities using the Quick Disabilities of the Arm, Shoulder and Hand (Quick DASH), which consists in eleven questions. 10 out of 11 eleven questions must be answered. All the answers are added and divided by the number of questions answered. Then, subtract 1 and multiply by 25. The higher the score, the greater the disability.
Upper Limb Lymphedema 27 (ULL-27) | Baseline and 5 weeks
  Quality of life in a questionnaire specific to patients with upper limb lymphedema secondary to breast cancer called Upper Limb Lymphedema 27 (ULL-27). The ULL-27 is a self-report questionnaire encompassing 27 questions with answers given on a 5-point Likert scale, ranging from "never" to "always" and is considered to measure the effects of lymphedema on health related quality of life. The questionnaire measures three domains: physical (15 items), psychological (7 items) and social (5 items), with scores ranging from 0 to 100 (100 being the best score possible).

CONTACTS AND LOCATIONS:
Overall Officials: María N Muñoz Alcaraz, Principal Investigator — Distrito Sanitario Córdoba Guadalquivir. Servicio Andaluz de Salud.; María V Olmo Carmona, Principal Investigator — UGC de Medicina Física y Rehabilitación IN. Hospital Universitario Reina Sofía; Antonio J Jiménez Vílchez, Principal Investigator — UGC de Medicina Física y Rehabilitación IN. Hospital Universitario Reina Sofía; Luis A Pérula de Torres, Principal Investigator — Unidad Docente de Medicina Familiar y Comunitaria de Córdoba; Jesús Serrano Merino, Principal Investigator — Distrito Sanitario Córdoba Guadalquivir. Servicio Andaluz de Salud.
Locations (1):
- Centro Periférico de Especialidades Castilla del Pino, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: Undecided
We are still developing the documents, we haven't decided yet if we are going to share them

REFERENCES:
- [Derived] Munoz-Alcaraz MN, Perula-de-Torres LA, Serrano-Merino J, Jimenez-Vilchez AJ, Olmo-Carmona MV, Munoz-Garcia MT, Bartolome-Moreno C, Olivan-Blazquez B, Magallon-Botaya R. Efficacy and efficiency of a new therapeutic approach based on activity-oriented proprioceptive antiedema therapy (TAPA) for edema reduction and improved occupational performance in the rehabilitation of breast cancer-related arm lymphedema in women: a controlled, randomized clinical trial. BMC Cancer. 2020 Nov 9;20(1):1074. doi: 10.1186/s12885-020-07558-x. PMID 33167921